CLINICAL TRIAL: NCT00394394
Title: Hydrochlorothiazide and Amiloride vs Hydrochlorothiazide and Enalapril: a Randomized Clinical Trial of Antihypertensive Effectiveness.
Brief Title: Antihypertensive Effectiveness of the Associations of Hydrochlorothiazide and Amiloride and Hydrochlorothiazide and Enalapril
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04002
Record Dates: First submitted 2006-10-30; First posted 2006-11-01 (Estimated); Last update posted 2006-11-01 (Estimated); Status verified 2006-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

INTERVENTIONS:
Drug: Amiloride 2,5/d or Enalapril/d 10 mg

SUMMARY:
The majority of hypertensive patients require antihypertensive associations to control their blood pressure. Most of clinical trials don't compare different associations using Hydrochlorothiazide 25 mg as the standard initial therapy and compare the associations using doses that are not equivalent.

This randomized trial where patients and investigators are blinded and compares the effectiveness two associations: Hydrochlorothiazide and Amiloride and Hydrochlorothiazide and Enalapril.

ELIGIBILITY:
Inclusion Criteria:

* patients who are using Hydrochlorothiazide 25mg/d at least in a four weeks treatment and had their office blood pressure not controlled (systolic or diastolic greater than 140 mmHg or 90 mmHg, respectively).

Exclusion Criteria:

* Established cardiovascular disease
* Diabetics in use of insulin
* Impairment renal in renal function
* Contraindications for the study medications

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-02

PRIMARY OUTCOMES:
Mean blood pressure measured with 24-hour ambulatory blood pressure monitoring after 12 weeks of follow-up

SECONDARY OUTCOMES:
Percentage of patients who needed to double the dose of enalapril or amiloride in forth or eighth week or use propranolol in the eighth week follow-up visiting.
Fasting blood glucose differences between the baseline and twelve-week follow-up visiting.
Serum potassium differences between the baseline and twelve-week follow-up visiting.
Serum total cholesterol, LDL- cholesterol, HDL- cholesterol and triglycerides differences between the baseline and twelve-week follow-up visiting.
Serum uric acid differences between the baseline and twelve-week follow-up visiting.
Urine microalbuminuria differences between the baseline and twelve-week follow-up visiting.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Gus, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Guerrero P, Fuchs FD, Moreira LM, Martins VM, Bertoluci C, Fuchs SC, Gus M. Blood pressure-lowering efficacy of amiloride versus enalapril as add-on drugs in patients with uncontrolled blood pressure receiving hydrochlorothiazide. Clin Exp Hypertens. 2008 Oct;30(7):553-64. doi: 10.1080/10641960802441906. PMID 18855259